CLINICAL TRIAL: NCT03699982
Title: Resting Energy Expenditure in Patients With Cystic Fibrosis: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left study institute.
Sponsor: CAMC Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-501
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystic fibrosis patients (Experimental): Patients with cystic fibrosis who are six year or older, who regularly receive care at the West Virginia University-Charleston Cystic Fibrosis Center, and agreed to participate in the study.
  Interventions: Other: Daily calorie target based on resting energy expenditure

INTERVENTIONS:
Other: Daily calorie target based on resting energy expenditure — Resting Energy Expenditure will be determined using the Harris-Benedict formula and indirect calorimetry testing. Additionally, a 48 Hour Dietary Recall will be completed to estimate approximate caloric intake at baseline.
  Participants will be instructed to increase their daily calorie intake based on the highest REE/caloric intake, whether by indirect calorimetry, the Harris-Benedict formula, or patient's estimated current caloric intake.

SUMMARY:
Cystic fibrosis is an inherited disorder that causes severe damage to the lungs, digestive system, and other organs in the body. Individuals with cystic fibrosis often have poor weight gain and growth that can negatively impact health further by worsening lung function. Additionally, persons with the disease typically need more than the usual calories on a daily basis.

Most institutions estimate these patients' caloric needs using weight, age, and sex based mathematical formulae. However, numerous studies show that use of these formulae often yields inaccurate caloric values. Use of indirect calorimetry may give more accurate estimates of caloric needs in patients with cystic fibrosis.

The aim of our study is to assess the accuracy of caloric estimates generated using one such widely used mathematical formula, the Harris-Benedict equation, and to compare this calorie value with that obtained from indirect calorimetry testing in pediatric and adult patients with cystic fibrosis.

Study investigators will use the newly calculated caloric requirements in dietary counseling. Changes in weight and lung function after 3 months will be compared to participants' historical changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis who are equal to or older than six years of age presenting to West Virginia University-Charleston Cystic Fibrosis Center for their regularly scheduled appointments/check-ups.
* Patients at the Cystic Fibrosis Center for at least 12 months.

Exclusion Criteria:

* Patients with cystic fibrosis who are younger than 6 years of age.
* Patients without cystic fibrosis.
* Patients currently pregnant.
* Cystic fibrosis patients with significant disease exacerbation (such as needing oral steroids or antibiotics, hospital admission within 30 days) or patients who currently having the flu or a serious upper respiratory infection.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure estimation | 1 hour
  Resting energy expenditure will be obtained using indirect calorimetry and the Harris-Benedict Equation.
Morphological variable changes | 3 months
  Weight/height/BMI changes after 3 months of intervention and historical weight/height/BMI changes occurring during the 12 preceding months (reported as 3 month means).
Changes in pulmonary function status | 3 months
  Changes in pulmonary function status, including FEV1%, after 3 months of intervention and historical pulmonary function status changes occurring during the 12 preceding months (reported as 3 month means).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dye, MD, Principal Investigator — CAMC and WVU-Charleston
Locations (1):
- CAMC - Women and Children's Hospital, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No